CLINICAL TRIAL: NCT02701881
Title: Comparison of the PrimAry Long Versus Short Coverage With Drug-Eluting Stents for Long FemoRopopliteal Artery DiseasE (PARADE II): Investigator-initiated Clinical Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2014-0072
Record Dates: First submitted 2016-02-29; First posted 2016-03-08 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Femoropopliteal Artery Disease
Keywords: Femoropopliteal Artery; Drug-eluting Stent; Endovascular Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Long stenting group (Experimental)
  Interventions: Device: Long stenting using drug-eluting stent (Zilver PTX)
- Short stenting group (Active Comparator)
  Interventions: Device: Spot stenting using drug-eluting stent (Zilver PTX)

INTERVENTIONS:
Device: Long stenting using drug-eluting stent (Zilver PTX) — Long stenting by full coverage of long femoropopliteal lesion with Zilver PTX after balloon angioplasty
  Arms: Long stenting group
Device: Spot stenting using drug-eluting stent (Zilver PTX) — Spot stenting by coverage of residual stenosis or flow-limiting dissection with Zilver PTX after balloon angioplasty of long femoropopliteal lesion
  Arms: Short stenting group

SUMMARY:
* Prospective, randomized, controlled, multi-center study
* A total of 220 subjects with long femoropopliteal lesions will be included according to inclusion and exclusion criteria.
* Patients will be randomized in a 1:1 manner into long stenting group versus short stenting group. and treated with Zilver PTX for long femoropopliteal lesions
* Patients will be followed clinically for 1 year after the procedure.
* Image study follow-up (Duplex US or CT angiography) will be performed at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Clinical criteria:

  1. Age 19 years of older
  2. Symptomatic peripheral artery disease:

     1. Moderate or severe claudication (Rutherford category 2 or 3)
     2. Critical limb ischemia (Rutherford category 4 or 5)
  3. Patients with signed informed consent
* Anatomical criteria:

  1. Target lesion length ≥150 mm by angiographic estimation
  2. Stenosis of more than 50% in femoropopliteal artery
  3. At least one patent (less than 50 percent stenosed) tibioperoneal runoff vessel.

Exclusion Criteria:

* A. Clinical criteria

  1. Acute critical limb ischemia
  2. Severe critical limb ischemia (Rutherford category 6)
  3. Major bleeding history within prior 2 months
  4. Known hypersensitivity or contraindication to any of the following medications: heparin, aspirin, clopidogrel or contrast agents
  5. Age > 85 years
  6. Severe hepatic dysfunction (> 3 times normal reference values)
  7. Significant renal dysfunction (Serum creatinine > 2.0 mg/dl
  8. Significant leucopenia, neutropenia, thrombocytopenia, anemia, or known bleeding diathesis
  9. LVEF(left ventricular ejection fraction) <40% or clinically overt congestive heart failure
  10. Pregnant women or women with potential childbearing
  11. Life expectancy <1 year due to comorbidity
* Angiographic criteria

  1. Previous bypass surgery or stenting of the superficial femoral artery
  2. Untreated inflow disease of the ipsilateral pelvic arteries (more than 50%stenosis or or occlusion
  3. Popliteal artery stenosis >50% at P2 or P3 segment

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2016-01; Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Primary patency rate | 12 months
  Absence of restenosis >50%

SECONDARY OUTCOMES:
Target vessel revascularization rate | 12 months
  repeat intervention or surgical treatment due to loss of patency at the target vessel

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Department of Internal Medicine, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park JI, Ko YG, Lee YJ, Lee SJ, Hong SJ, Ahn CM, Kim JS, Kim BK, Hong MK, Yu CW, Rha SW, Park JK, Min PK, Yoon CH, Lee SR, Park SH, Choi DH. Long coverage with drug-eluting stents is superior to spot coverage for long femoropopliteal artery disease: PARADE II study. Front Cardiovasc Med. 2022 Oct 19;9:1022071. doi: 10.3389/fcvm.2022.1022071. eCollection 2022. PMID 36337904